CLINICAL TRIAL: NCT04528706
Title: An Open-label, Multicenter Study in Male Pediatric Patients With Cerebral X-linked Adrenoleukodystrophy (Cald) to Assess the Effects of MIN-102 Treatment on Disease Progression Prior to Human Stem Cell Transplant (HSCT)
Brief Title: A Clinical Study in Male Pediatric Patients With Cerebral X-linked Adrenoleukodystrophy (Cald) to Assess the Effects of MIN-102 Treatment on Disease Progression Prior to Human Stem Cell Transplant (HSCT)
Acronym: NEXUS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Minoryx Therapeutics, S.L. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT-2-02
Record Dates: First submitted 2020-07-31; First posted 2020-08-27 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-01

CONDITIONS: Cerebral Adrenoleukodystrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MIN-102 (Experimental)
  Interventions: Drug: MIN-102

INTERVENTIONS:
Drug: MIN-102 — Once-daily dosing with a volume specified by the pharmacokineteic specialist to achive the desired plasma exposure. Min-102 Oral suspension, strength 15mg/ml.

SUMMARY:
An Open-Label, multicenter study in male pediatric patients with cerebral x-linked adrenoleukodystrophy (cald) to assess the effects of MIN-102 treatment on disease progression prior to human stem cell transplant (HSCT)

ELIGIBILITY:
Inclusion Criteria:

* Males aged ≥2 and ≤12 years with a diagnosis of X-linked ALD
* White matter involvement as determined by cerebral MRI lesions without Gd enhancement at baseline (Population 1), or with Gd enhancement at baseline (Population 2).
* Major Functional Disabilities (MFD) score of 0.
* Baseline Loes score >0 and ≤10
* Gadolinium Intensity Score >2

Exclusion Criteria:

* Previous HSCT
* Too far progressed inflammatory brain lesions

Ages: 2 Years to 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Estimated)
Dates: Start 2019-09-13 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
evaluate whether MIN-102 can halt disease progression of cALD if administered prior to hematopoietic stem-cell transplantation (HSCT), as determined by serial clinical and MRI investigations in pediatric subjects. | 6 months- 2 years
"arrested disease" will be assessed at 24 weeks and at 96 weeks | at 24 weeks and 96 weeks
  arrested disease is defined using: Cahnge in NFS from Baseline, Free of MFD and lack of lesion progression on MRI

CONTACTS AND LOCATIONS:
Locations (5):
- Hernan Amartino, Bueno Aires, Buenos Aires, Argentina
- CHU Kremlin Bicêtre, Paris, France
- Germany (2):
  - Universitätsmedizin Göttingen Georg-August-Universität, Göttingen
  - Universitätsklinikum Hamburg-Eppendorf Klinik und Poliklinik für Kinder- und Jugendmedizin, Hamburg
- Hospital Sant Joan de Déu, Barcelona, Spain